CLINICAL TRIAL: NCT00100308
Title: Unfractioned Heparin for Treatment of Sepsis: A Randomized Clinical Trial (The HETRASE Study)
Brief Title: Unfractioned Heparin for Treatment of Sepsis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government)
Responsible Party: Fabian Jaimes MD.,MSc., PhD, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COLCIENCIAS -11150416347
Record Dates: First submitted 2004-12-28; First posted 2004-12-29 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Sepsis; Bacterial Infections
Keywords: sepsis; Randomized clinical trial; Heparin; Therapy
MeSH Terms: conditions — Sepsis; Bacterial Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Standard treatment plus unfractioned heparin low-dose continuous infusion
  Interventions: Drug: Unfractioned heparin
- 2 (Placebo Comparator): Standard treatment plus placebo
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Unfractioned heparin — Low-dose continuous-infusion, 500 units/hour per seven days
  Arms: 1
Drug: saline — Saline placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether low dose continuous infusion of unfractioned heparin (500 units/hour), in addition to the standard treatment, is efficacious as complementary therapy for sepsis patients.

DETAILED DESCRIPTION:
Sepsis is considered a leading cause of death worldwide with approximately 18 million cases annually and a mortality rate of almost 30%. The search for efficacious therapeutic approaches has largely failed and only a few of the recent interventions, such as activated protein C and low dose steroids, have shown some success in improving survival. However, these interventions were tested only in patients with severe sepsis and/or septic shock and although these groups exhibit the highest mortality, they represent less than 50% of the total affected population. Furthermore, these interventions necessitate special devices, tests and/or drugs that might be unavailable or simply unaffordable in resource-limited settings.

Animal and human models have suggested that heparin, in addition to successfully inhibiting the coagulation cascade, may also modulate the wide array of responses to infection. Furthermore, the three clinical trials for recombinant anticoagulants allowed the use of prophylactic treatment for venous thrombosis with a dose of unfractioned heparin (UFH) of up to 10,000 or 15,000 units subcutaneously per day. When those who did receive heparin were compared to those who did not in the placebo arms of the clinical trials, all three studies showed a higher mortality in the subgroups that did not receive heparin. Although this is not a randomized comparison, a constant result in three different study populations with variable entry criteria, along with the natural heterogeneity of the illness, strongly fosters the hypothesis that heparin might reduce, beyond its known anticoagulant and antithrombotic properties, the overall mortality for sepsis.

In this project, we propose a phase II/III, randomized, double-masked, placebo-controlled, single-center clinical trial with a total sample size of 310 patients, for testing low dose continuous infusions of UFH (500 units/hour) for 7 days, as complementary treatment for septic patients. Our primary aims are to estimate the effects of UFH on length of stay and change from baseline Multiple Organic Dysfunction (MOD) score. Secondary objectives are to estimate the effects of UFH on 28-day all-cause mortality, and to estimate the possible effect-modification on 28-day all-cause mortality, in subgroups defined by site of infection and baseline values of APACHE II score, MOD score and D-dimer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an infection defined by clinical and/or microbiological criteria in accordance with modified CDC definitions for nosocomial infections
* Patients must present with one or more of the GENERAL VARIABLES, AND one or more of the INFLAMMATORY VARIABLES within 24 hours before admission to the study

GENERAL VARIABLES:

* Temperature (oral or axillary) > 38ºC or < 36ºC,
* Heart rate > 90 beats/min,
* Respiratory rate > 20 breaths/min,
* Altered mental status determined by Glasgow Coma Scale < 15,
* Systolic blood pressure < 90 mm Hg or a decrease > 40 mm Hg

INFLAMMATORY VARIABLES:

* WBC > 12,000 μL-1 or < 4,000 μL-1 or with > 10% immature forms,
* Plasma C-reactive protein > 5 mg/dL.

These variables should not be attributable to an underlying disease other than infection or due to the effects of concomitant therapy.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Platelet count < 60,000/mm3.
* Increased risk for bleeding: * Any patient who has undergone major surgery, defined as surgery that required general or spinal anesthesia, performed within the 12-hour period immediately preceding admission to the hospital; any postoperative patient who demonstrates evidence of active bleeding; or any patient with planned or anticipated major surgery during the first 12 hours after admission to the hospital. * History of: severe head trauma that required hospitalization, intracranial surgery, or stroke within 3 months of study entry; or any history of intracerebral arteriovenous malformation, cerebral aneurysm, or central nervous system mass lesion. * History of congenital bleeding diatheses, such as hemophilia. * Gastrointestinal bleeding within 6 weeks of study entry that required medical intervention unless definitive surgery has been performed. * Trauma patients at increased risk of bleeding, for example: flail chest; significant contusion to lung, liver, or spleen; retroperitoneal bleed; pelvic fracture; or compartment syndrome.
* Patients with a known hypercoagulable condition including activated Protein C resistance; a hereditary deficiency of Protein C, Protein S, or antithrombin; presence of anticardiolipin antibody, antiphospholipid syndrome, lupus anticoagulant or homocysteinemia; or patients with a recently documented (within 3 months of study entry) or highly suspected deep venous thrombosis or pulmonary embolism.
* Patients taking or requiring the following medications: * Therapeutic heparin, defined as UFH dosed to treat an active thrombotic or embolic event within the 12 hours prior to study entry or LMWH used at any dose higher or more frequent than the recommended dose on the product label for prophylaxis within the 12 hours prior to study entry. * Warfarin, if used within 7 days of study entry. * Thrombolytic treatment within 3 days of study entry (for example, streptokinase, rtPA, and urokinase). * Glycoprotein IIb/IIIa antagonists within 7 days of study entry.
* Patients with known esophageal varices, chronic jaundice, cirrhosis, or chronic ascites.
* Patients not expected to survive 28 days given their preexisting, uncorrectable medical condition. This criterion includes patients with, or suspected to have, poorly controlled neoplasms or other end-stage processes, such as end-stage cardiac disease, prior cardiac arrest, end-stage lung disease, or end-stage liver disease.
* Patients with chronic renal failure on either hemodialysis or peritoneal dialysis.
* HIV positive patients with most recent CD4 count < 200/mm3.
* Patients who have undergone bone marrow, liver, lung, kidney or pancreas transplantation.
* Inability or unwillingness of patients or legal representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline Multiple Organ Dysfunction (MOD) score | 15 days
Length of stay | During hospitalization

SECONDARY OUTCOMES:
28-day all-cause mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Fabián A Jaimes, MD, MSc, PhD, Principal Investigator — Universidad de Antioquia
Locations (1):
- Hospital Universitario San Vicente de Paul, Medellín, Antioquia, Colombia